CLINICAL TRIAL: NCT06601972
Title: Clinical and Radiographic Evaluation of Partial Caries Removal in Permanent Molars Restored Using Giomer Compared to Resin Composite Restorations After 24 Months (A Randomized Clinical Trial)
Brief Title: Partial Caries Removal in Permanent Molars Restored Using Giomer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NewGiza University (Other)
Responsible Party: Principal Investigator, Omar Shaalan, Associate professor of conservative dentistry, NewGiza University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: giomervscomp
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Caries, Dental
Keywords: partial caries removal; bioactive; giomer
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Giomer (Experimental): Low-shrinkage bioactive material
  Interventions: Procedure: Beautifil II LS (Low-Shrinkage)
- Nanohybrid composite (Active Comparator): Universal Nano-hybrid composite
  Interventions: Procedure: Nanohybrid resin composite

INTERVENTIONS:
Procedure: Beautifil II LS (Low-Shrinkage) — The most remarkable feature of this light-cured universal composite for anterior and posterior restorations is its unique shrinkage of 0.85 percent by volume
  Arms: Giomer
Procedure: Nanohybrid resin composite — Nanohybrid resin composites are the most popular, because they improve the distribution of fillers in the matrix by combining nanoparticles with submicron particles to achieve better mechanical, chemical, and optical properties
  Arms: Nanohybrid composite

SUMMARY:
Dental manufacturers' constant tweaks and improvements to composite compositions have resulted in a wider spectrum of restorative materials with positive long-term clinical performance. For example, the creation of bioactive giomer material with proven continuous multi-ion release has been beneficial in avoiding demineralization and imparting acid resistance to enamel and dentin.

DETAILED DESCRIPTION:
Giomer resin not only reduces the risk of secondary caries around restorations by releasing fluoride ions, but it also has good esthetic, physical, and handling features. Furthermore, advancements have been made to reduce giomer resin polymerization shrinkage by incorporating filler technology into the matrix system. As a result of these efforts, giomer resin is currently distinguished by its low shrinkage feature. According to the manufacturer, low shrinkage giomer resin has volumetric shrinkage of 0.8% and a polymerization shrinkage stress of 2.72 MPa. Several investigations were carried out to examine the overall clinical performance of low shrinkage giomer resin with equivalent success rates when compared to other restorative materials. The aim of the current study is to evaluate the effect of giomer in maintaining pulp health and dentin bridge formation after partial caries removal in permanent teeth with deep occlusal carious lesion when compared to resin composite restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria of participants:

   * 18 -35 years.
   * Not received antibiotic therapy since 1 month before sampling.
   * Males or Females (Both genders).
   * Co-operative patients approving the trial.
   * Good to fair oral hygiene
2. Inclusion criteria of teeth:

   * Class I cavitated lesions in permanent molars (reaching >1/2 of the dentin on radiographic examination)
   * Absence of spontaneous pain; negative sensitivity to percussion; and absence of periapical lesions (radiographic examination).

Exclusion Criteria:

1. Exclusion criteria of participants:

   * known allergic reaction to resinous materials.
   * Systemic disease or severe medical complications.
   * Periodontal problem.
   * Bruxism
   * Poor oral hygiene
2. Exclusion criteria of teeth:

   * Class II caries lesion
   * Shallow or enamel caries
   * Teeth with periapical lesions.
   * Mobile teeth, arrest caries and non-vital teeth

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | From enrollment to the end of treatment at 24 months
  The primary outcome of the present clinical trial is success rate, expressed as a binary variable indicating whether the restored tooth maintained its pulp vitality after 24 months. Success will be evaluated by a positive response to cold pulp testing, absence of spontaneous pain, no tenderness to percussion, absence of periapical radiolucency.

SECONDARY OUTCOMES:
Dentin bridge formation | From enrollment to the end of treatment at 24 months
  Dentin bridge formation will be evaluated by digital radiographs taken with standardized exposure parameters according to standardized procedure by placement of film holders in paralleling technique. Dentin bridge formation will be measured by millimeters (mm)

IPD SHARING:
Plan to Share IPD: No
confidentiality, risk of data misinterpretation